CLINICAL TRIAL: NCT05720312
Title: A Preliminary Investigation of Two Repetitive Transcranial Magnetic Stimulation (rTMS) Strategies to Treat Cannabis Use Disorder
Brief Title: Investigating Two rTMS Strategies to Treat Cannabis Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Daniel McCalley, Postdoctoral Scholar, Psychiatry, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 68235
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cannabis Use Disorder
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dorsolateral Prefrontal Cortex (DLPFC) (Experimental): 36 sessions of high frequency (10Hz) rTMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Ventromedial Prefrontal Cortex (vmPFC) (Experimental): 36 sessions of low frequency (1Hz) rTMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Patterned pulsed magnetic stimulation delivered using an electromagnet. We will use a MagVenture rTMS device and a Cool-B65 coil.

SUMMARY:
In this trial we will work with a group of participants who are having problems related to marijuana use (they have Cannabis Use Disorder) and who want to reduce the amount of marijuana they use or quit using marijuana completely. We are testing to see if a treatment called repetitive transcranial magnetic stimulation (rTMS) can help them achieve that goal when combined with a brief three-session counseling therapy. Participants will receive rTMS to one of two different parts of the brain (the dorsolateral prefrontal cortex--the DLPFC or the ventromedial prefrontal cortex--the vmPFC) to see if applying rTMS to one brain area is more helpful than the other brain area.

DETAILED DESCRIPTION:
In this preliminary trial, we will test whether applying repetitive transcranial magnetic stimulation (rTMS) to one of two brain areas will help participants with Cannabis Use Disorder reduce the amount of cannabis they use or quit using cannabis completely. To do so, we will recruit participants from the community (or addictions medicine treatment centers) who meet the criteria for Cannabis Use Disorder (heavy use of cannabis causing social, occupational, or health problems) and want to either substantially reduce the amount of cannabis they use or quit using cannabis entirely. Participants will be randomized (in a 1:1 allocation) to receive rTMS to either the left dorsolateral prefrontal cortex (DLPFC) or the ventromedial prefrontal cortex (vmPFC). All participants will also receive evidence-based counseling to help them reduce the amount of cannabis they use. We will deliver study treatment with rTMS to participants over 18-study-visits occurring either two or three times each week and then will see whether the study treatment has helped by meeting with participants four times over six weeks. We will also see how the rTMS effected brain function by having participants undergo two scans using magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Participants must be between the ages of 18 and 60.
3. Participants must meet DSM-5 criteria for at least moderate Cannabis Use Disorder, with use of at least 20 out of the last 28 days.
4. Participants must express a desire to reduce cannabis use or quit.
5. Participants must have a positive UDS for cannabis during their enrollment visit (confirming they are regular users).
6. The investigative team must believe each participant is a good study-candidate.

Exclusion Criteria:

1. Participants must not be pregnant or breastfeeding.
2. Participants must not meet moderate or severe use disorder of any other substance with the exception of tobacco/nicotine.
3. Participants must not be on any medications that have central nervous system effects that have changed in the past 4-weeks.
4. Participants must not have a history of/or current psychotic disorder or bipolar disorder.
5. Participants must not have any other Axis I condition requiring current treatment.
6. Participants must not have a history of Dementia or other cognitive impairment.
7. Participants must not have active suicidal ideation, or a suicide attempt within the past 180 days.
8. Participants must not have any contraindications to receiving rTMS or MRI (e.g. metal implanted above the head, history of seizure, any known brain lesion).
9. Participants must not have any unstable general medical conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sahlem, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants receive 6 to 9 weeks of active treatment, then enter a 7 week follow-up period, from the last treatment (up to 1 week) plus 6 weeks post-treatment.
Pre-assignment Details: 22 participants signed informed consent, and 20 were randomized to treatment.
Groups:
- Dorsolateral Prefrontal Cortex (DLPFC): 36 sessions of high frequency (10Hz) repetitive Transcranial Magnetic Stimulation (rTMS).
Period: Treatment Period (6 to 9 Weeks)
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Ventromedial Prefrontal Cortex (vmPFC)
Started | 10 | 10
Completed | 8 | 8
Not Completed | 2 | 2
Period: Follow-up Period (6 Weeks)
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Ventromedial Prefrontal Cortex (vmPFC)
Started | 8 | 8
Completed | 6 | 8
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Ventromedial Prefrontal Cortex (vmPFC) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (6.5) | 37.7 (10.8) | 33.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 3 | 4
  White | 0 | 3 | 3
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number (%) of Participants Who Started and Completed Treatment
Time Frame: 6 to 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Ventromedial Prefrontal Cortex (vmPFC)
Number analyzed (Participants) | 10 | 10
Participants | 8 | 8

2. Primary Outcome: Number (%) of Participants Who Had Successful Generation of Functional Magnetic Resonance Imaging (fMRI) Targets
Time Frame: Day 1 (90 minutes to complete scan)
Measure: Count of Participants; unit: Participants
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Ventromedial Prefrontal Cortex (vmPFC)
Number analyzed (Participants) | 10 | 10
Participants | 10 | 9

3. Primary Outcome: Number (%) Weeks of Abstinence From Cannabis
Description: Number (%) of weeks where the participant does not use any cannabis.
Time Frame: 13 weeks (final 7 weeks of active treatment plus 6-week post-treatment follow-up)
Measure: Count of Units; unit: patient weeks
Units Other Than Participants: patient weeks
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Ventromedial Prefrontal Cortex (vmPFC)
Number analyzed (Participants) | 10 | 10
Number analyzed (patient weeks) | 130 | 130
patient weeks | 0 | 56

4. Secondary Outcome: Number of Days of Use Per Week.
Description: Number of days per week (0-7) where the participant uses any cannabis. At the time of enrollment participants were asked to recall the number of days of cannabis use per week for the 4 weeks prior to enrollment. Participants were then asked (over a period of 7 weeks) to recall days of use at the last fMRI visit (during prior week) and at the week 2, 4, and 6 follow-up visits. Average values are reported for the 4-week period prior to enrollment and the 7-week period at end of treatment at follow-up.
Time Frame: 4 weeks prior to baseline assessment and 7 weeks at the end of treatment through 6-week post-treatment follow-up
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Ventromedial Prefrontal Cortex (vmPFC)
Number analyzed (Participants) | 10 | 10
days per week
  Baseline assessment | 6.82 (0.38) | 6.68 (0.69)
  End of treatment / Follow-up | 5.27 (1.95) | 2.82 (3.25)

5. Secondary Outcome: Average Number of Use Sessions Per Week.
Description: Number of use sessions per week where the participant uses any cannabis. At the time of enrollment participants were asked to recall the number of cannabis use sessions per week for the 4 weeks prior to enrollment. Participants were then asked (over a period of 7 weeks) to recall the number of cannabis use sessions at the last fMRI visit (during prior week) and at the week 2, 4, and 6 follow-up visits. Average values are reported for the 4-week period prior to enrollment and the 7-week period at end of treatment at follow-up.
Time Frame: 4 weeks prior to baseline assessment and 7 weeks at the end of treatment through 6-week post-treatment follow-up
Measure: Mean (Standard Deviation); unit: use sessions per week
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Ventromedial Prefrontal Cortex (vmPFC)
Number analyzed (Participants) | 10 | 10
use sessions per week
  Baseline assessment | 50.33 (27.28) | 32.55 (18.52)
  End of treatment / Follow-up | 29.68 (27.26) | 11.69 (18.71)

6. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) Scale Score
Description: The Q-LES-Q-SF overall score range is from 14 to 70, with higher scores indicating greater satisfaction and enjoyment. The total score is expressed as a percentage of the maximum possible score (1-100).
Time Frame: Baseline and end of the follow-up period (12 to 15 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Ventromedial Prefrontal Cortex (vmPFC)
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline assessment | 56.25 (13.61) | 54.82 (11.97)
  End 6-week follow-up | 62.50 (11.01) | 67.63 (11.15)

7. Secondary Outcome: Number of Participants Who Had a Period of 4-consecutive Weeks of Abstinence During the Follow-up Period
Description: Based on patient self-report of any 4-week period of abstinence
Time Frame: Follow-up period (final week of active treatment plus 6-week post-treatment follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | Dorsolateral Prefrontal Cortex (DLPFC) | Ventromedial Prefrontal Cortex (vmPFC)
Number analyzed (Participants) | 10 | 10
Participants | 0 | 4

ADVERSE EVENTS:
Time Frame: Up to 15 weeks (6 to 9 weeks of treatment plus 6 week follow up)
Groups:
- DLPFC - Treatment Period; DLPFC - Follow-up Period: 36 sessions of high frequency (10Hz) rTMS.
- vmPFC - Treatment Period; vmPFC - Follow-up Period: 36 sessions of low frequency (1Hz) rTMS.
Arm/Group | DLPFC - Treatment Period | vmPFC - Treatment Period | DLPFC - Follow-up Period | vmPFC - Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/10 | 4/10 | 0/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DLPFC - Treatment Period (N=10) | vmPFC - Treatment Period (N=10) | DLPFC - Follow-up Period (N=8) | vmPFC - Follow-up Period (N=8)
Fatigue (General disorders) | 2 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 0
Transient Vision Change (Eye disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT05720312/Prot_SAP_000.pdf